CLINICAL TRIAL: NCT03329222
Title: A Randomised, Double Blind, Controlled, Multi-centre Study to Assess the Efficacy of an Infant Formula in the Dietary Management of Infantile Colic
Brief Title: An Infant Formula Trial on Dietary Management of Infantile Colic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: National University Hospital, Singapore (Other); Phramongkutklao College of Medicine and Hospital (Other); Maharaj Nakorn Chiang Mai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: EBB16SI06749
Record Dates: First submitted 2017-10-03; First posted 2017-11-01 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: Randomized, two arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): An infant formula which contains specific hydrolysed proteins with a fat blend, prebiotics mixture, starch and reduced lactose
  Interventions: Other: Specific hydrolysed proteins
- Control group (Active Comparator): Standard cow's milk with prebiotics mixture
  Interventions: Other: Standard cow's milk with prebiotics mixture

INTERVENTIONS:
Other: Specific hydrolysed proteins — An infant formula which contains specific hydrolysed proteins with a fat blend, prebiotics mixture, starch and reduced lactose
  Arms: Intervention group
Other: Standard cow's milk with prebiotics mixture — Standard cow's milk with prebiotics mixture
  Arms: Control group

SUMMARY:
A randomised, double blind, controlled, multi-centre study to assess the efficacy of an infant formula in the dietary management of infantile colic.

DETAILED DESCRIPTION:
A randomised, double blind, controlled, multi-centre study to assess the efficacy of an infant formula in the dietary management of infantile colic.

The hypothesis of the study is that the test product, compared to the control formula, will reduce the crying time in infants with infantile colic.

The various time points of the outcome are:

V1 (screening : Day -5 to day 0); V2 ( Randomization: Day 0); V3 (Day 7); V4 (Day 21); Phone Call (Day 28); V5 (End -intervention: Day 42); V6 (Day 56)

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 21-56 days (both inclusive);
2. Gestation age 37-42 weeks;
3. Normal birth weight for gestational age and gender
4. 5-minute APGAR score >7;
5. Diagnosed with infantile colic ;
6. Fully formula fed for at least 7 days before randomisation;
7. Written informed consent from the parent and/or legal representative.

Exclusion Criteria:

1. Any plausible cause of inconsolable crying as judged by the investigator;
2. Presence of non-functional vomiting or failure to thrive;
3. Presence of any congenital defects in the gastrointestinal system or other defects preventing oral nutrition;
4. Congenital condition and/or previous or current illness/infection and (or) medication use that could interfere with the main study outcomes;
5. Known cow's milk protein allergy, lactose intolerance, or galactosaemia; including presence of any allergic manifestations;
6. Received any special formula (e.g. lactose-free, hydrolysed protein);
7. Received any of the following products/medication within 7 days before randomisation:

   1. Probiotics
   2. Systemic antibiotics
   3. Prokinetics
   4. Proton pump inhibitors
8. Twins or triplets or other infant(s) <6 months of age living in the same household;
9. Incapability of the parent(s) to comply with the study protocol or investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements;
10. Current participation in another clinical study involving investigational or marketed products.

Ages: 21 Days to 56 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Daily inconsolable crying time using data recorded on subject's diaries | 6 weeks
  Daily inconsolable crying time over 6 weeks

SECONDARY OUTCOMES:
Daily crying time using data recorded on subject's diaries | 6 weeks
  Daily crying time over 6 weeks of intervention
Daily fussing time using data recorded on subject's diaries | 6 weeks
  Daily fussing time over 6 weeks of intervention
Daily inconsolable fussing time using data recorded on subject's diaries | 6 weeks
  Daily inconsolable fussing time over 6 weeks of intervention
Daily stool frequency using data recorded on subject's diaries | 6 weeks
  Daily stool frequency over 6 weeks of intervention
Daily stool consistency using data recorded on subject's diaries | 6 weeks
  Daily stool consistency over 6 weeks of intervention
The frequency of subject's GI symptoms of digestion in the 7-day period prior to the visit using the Infant gastrointestinal symptoms questionnaire | 6 weeks
  Gastrointestinal symptoms using the Infant gastrointestinal symptoms questionnaire during the 6-week intervention period
The intensity of subject's GI symptoms of digestion in the 7-day period prior to the visit using the Infant gastrointestinal symptoms questionnaire | 6 weeks
  Gastrointestinal symptoms using the Infant gastrointestinal symptoms questionnaire during the 6-week intervention period

CONTACTS AND LOCATIONS:
Locations (2):
- National University Hospital, Singapore, Singapore, Singapore
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No